CLINICAL TRIAL: NCT06191289
Title: Clarifying the Endocrinology of Acute Risk 4 (CLEAR-4): Neurocognitive Mechanisms of Perimenstrual Estrogen Effects on Suicidality
Brief Title: Neurocognitive Mechanisms of Perimenstrual Estrogen Effects on Suicidality
Acronym: CLEAR-4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding changes necessitated the preliminary conclusion of the study; it will be used for feasibility data.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tory Anne Eisenlohr-Moul, Associate Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-1560
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: MENSTRUAL CYCLE; HORMONES; ESTROGEN; REWARD; EXECUTIVE FUNCTION
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Crossover 2-condition placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transdermal Estradiol (Experimental): .1mg per 24 hours transdermal estradiol applied to the skin weekly, for 14 days.
  Interventions: Drug: Transdermal Estradiol
- Placebo (Placebo Comparator): Clear patch manufactured to mimic the E2 patch applied to the skin weekly, for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Transdermal Estradiol — 1mg/24hr transdermal estradiol for 14 days starting day 7 after positive urine luteinizing hormone test
  Other Names:
  Climara
  Arms: Transdermal Estradiol
Other: Placebo — Weekly application of a placebo patch for 14 days starting day 7 after positive urine luteinizing hormone test
  Arms: Placebo

SUMMARY:
This within-person, crossover, 2-condition, placebo-controlled study compares the impact of two perimenstrual conditions on severity of suicidal symptoms in females with past-month suicidality but minimal risk of imminent suicide attempt. The two conditions are (1) perimenstrual administration of estradiol and (2) natural perimenstrual withdrawal from estradiol during placebo.

DETAILED DESCRIPTION:
Previous work from our group demonstrates that perimenstrual worsening of suicidal thoughts in females is caused by normal perimenstrual withdrawal from the ovarian steroid estradiol (E2), since perimenstrual administration of E2+P4 or E2 alone prevented the perimenstrual worsening of suicidal ideation observed under placebo. In the present study, we follow up on that work with an additional mechanistic crossover trial in which E2 will be administered perimenstrually (E2 condition) or not (PBO condition) and neurocognitive mechanisms of suicidal symptom improvement will be probed.

50 (30 completers) female outpatients, with past-month suicidal ideation but minimal imminent risk for attempt, will complete self-reports and clinical interviews measuring the presence and severity of suicidal ideation in each of two conditions (A, B: order randomized across two menstrual cycles): (A) perimenstrual E2 withdrawal/depletion (under placebo), (B) perimenstrual administration of E2. A washout cycle will separate conditions. Analyses will compare the perimenstrual trajectories of symptoms and suicidality across the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adhere to medication regimen
* Speaks English
* Assigned female at birth with intact ovaries
* Premenopausal
* Normal menstrual cycles between 24-32 days
* Under current care of an outpatient mental health provider with visits occurring at least once every 3 months.
* At least 1 year postpartum.
* Willing to use a barrier method of birth control during the study.
* Normal weight (BMI between 18-29)
* Must report at least some recent suicidal ideation (in the past month) at the time of recruitment.
* Must be categorized as having acceptably low imminent risk for suicidal crisis/attempt by a licensed clinical psychologist utilizing evidence-based clinical and research guidelines for imminent suicide risk management.

Exclusion Criteria:

* Must not be pregnant, breastfeeding, or trying to become pregnant.
* Must not be taking any form of exogenous hormones or hormonal intrauterine device, and must have ended previous use of hormonal preparations at least one month prior to the study.
* Must not have a personal history of any chronic medical condition, including but not limited to metabolic or autoimmune disease, epilepsy, endometriosis, cancer, diabetes, cardiovascular, gastrointestinal, hepatic, renal, or pulmonary disease, and no personal or first degree family history of thromboembolic events.
* Any current cigarette smoking is exclusionary.
* Must not report a history of clinical diagnosis or treatment for postpartum depression or premenstrual dysphoric disorder (Note: Premenstrual Dysphoric - - - Disorder diagnosis must have been made based on prospective daily ratings).
* Must not report any history of manic episode, any history of psychotic symptoms, or current substance use disorder.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-03-16 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Early-Luteal-to-Perimenstrual Worsening of Daily Passive Suicidal Ideation (PSI) | Mean daily rating in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean daily rating in the early luteal phase (Days +2, +3, +4, +5, and +6
  Three daily survey questions assessing PSI will be administered each day (i.e., "I wished I were dead", "I wish I could go to sleep and not wake up", "I thought that life was not worth living"; scale from 1 (Not at All) to 5 (Extremely)). Composite mean scores for these 3 items are computed, providing a single number for each day, with higher daily values representing more severe PSI.
  Early-luteal-to-perimenstrual worsening of daily PSI is estimated for each person in each condition as the mean of scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0).
Early-Luteal-to-Perimenstrual Worsening of Daily Active Suicidal Ideation (ASI) | Mean daily rating in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean daily rating in the early luteal phase (Days +2, +3, +4, +5, and +6
  Three daily survey questions assessing ASI will be administered each day (i.e., "I thought about killing myself", "I wanted to kill myself", "I had the urge to kill myself"; scale from 1 (Not at All) to 5 (Extremely)). Composite mean scores for these 3 items are computed, providing a single number for each day, with higher daily values representing more severe ASI.
  Early-luteal-to-perimenstrual worsening of daily ASI is estimated for each person in each condition as the mean of scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0).
Early-Luteal-to-Perimenstrual Increase in the Probability of Daily Suicidal Planning (SP) | Mean daily dichotomous outcome (ranging from 0-1) in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean in the early luteal phase (Days +2,
  Two questions from the ASIQ assessing SP will be administered each day in an adapted daily format (i.e., "I thought about how I might kill myself", "I thought about when I might kill myself"; scale from 1 (Not at All) to 5 (Extremely)). Daily dichotomous scores will be derived such that if either of these two items are endorsed with a score higher than 1 (not at all) on a given day, the composite score will be 1 (otherwise the score will be 0) for that day.
  Early-luteal-to-perimenstrual increase in the probability of daily SP is estimated for each person in each condition as the mean of dichotomous daily scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean of dichotomous scores in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0).

SECONDARY OUTCOMES:
Perimenstrual Reward Positivity (RewP) | Mean RewP amplitude in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline)
  The reward positivity (RewP), measured with electroencephalography, is an event-related potential (ERP) component index of neural responsiveness to receipt of reward. Approximately 300 milliseconds (ms) after computerized task feedback indicating monetary reward, the ERP at frontocentral recording sites is characterized by a relative positivity; an apparent negativity is observed following feedback indicating monetary loss. The relative difference in ERP amplitudes in response to reward as compared to loss is referred to as the Reward Positivity. During each experimental perimenstrual phase (E2 vs. placebo), participants will participate in a gambling task while EEG is used to record the averaged RewP amplitude.
Early-Luteal-to-Perimenstrual Worsening of daily self-reported anhedonia | Mean daily rating in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean daily rating in the early luteal phase (Days +2, +3, +4, +5, and +6
  Three daily items assessing anhedonia will be administered each day (i.e., "Didn't enjoy things", "Had less interest in things", and "Felt unmotivated to do things"; scale from 1 (Not at All) to 6 (Extreme)). Composite mean scores for these 3 items are computed for each day, providing a single number for each day, with higher daily values representing more anhedonia.
  Early-luteal-to-perimenstrual worsening of daily anhedonia is estimated for each person in each condition as the mean of scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0).
Early-Luteal-to-Perimenstrual change (improvement) in daily N-Back performance | Mean daily rating in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean daily rating in the early luteal phase (Days +2, +3, +4, +5, and +6
  Participants will complete a daily at-home working memory computerized task: the N-Back task. Number of "hits" (i.e., correctly indicated targets) in this task will serve as our measure of daily working memory behavioral performance, with higher daily values representing better working memory performance.
  Early-luteal-to-perimenstrual change (calculated as improvement) of daily N-Back scores is estimated for each person in each condition as the mean of scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0). Therefore, positive values represent a perimenstrual improvement in working memory performance, and negative values represent a perimenstrual worsening.
Early-Luteal-to-Perimenstrual Worsening of daily self-reported working memory failures (WMF) | Mean daily rating in the perimenstrual phase (Days -3, -2, -1, and +1 relative to menses onset where menses onset is day +1 and there is no 0 on the menses-onset timeline) minus the mean daily rating in the early luteal phase (Days +2, +3, +4, +5, and +6
  Three questions assessing WMF will be administered each day (i.e., "Had difficulty concentrating", "I forgot things", and "I got distracted easily"; scale from 1 (Not at All) to 6 (Extreme)). Composite mean scores for these 3 items are computed daily, providing a single number for each day, with higher daily values representing more severe WMF.
  Early-luteal-to-perimenstrual worsening of WMF is estimated for each person in each condition as the mean of scores in the perimenstrual phase (Days -3 to +1 relative to menses onset) minus the mean in the early luteal phase (Days +2 to +6 relative to the luteinizing hormone surge at day 0).

CONTACTS AND LOCATIONS:
Overall Officials: Tory A Eisenlohr-Moul, Ph.D., Principal Investigator — University of Illinois at Chicago; Elizabeth Mulligan, Ph.D., Principal Investigator — University of Illinois at Chicago; Katja M Schmalenberger, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Neuropsychiatric Institute, Chicago, Illinois, United States